CLINICAL TRIAL: NCT06978140
Title: Decisions During Drinking: Phase 3 Feasibility Study
Brief Title: Decisions During Drinking
Acronym: D3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Brittney Hultgren, Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00021311; K01AA027771-05 (NIH)
Record Dates: First submitted 2025-04-16; First posted 2025-05-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Alcohol
Keywords: alcohol-related consequences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D3 online health information and text-messages (Experimental): Participants receiver personalized health information feedback across 5-7 online modules over 20-30 days along with text-message health information
  Interventions: Behavioral: Personalized feedback
- Assessment only control (No Intervention): Participants will receive questionnaires similar to intervention group but will not receive any health information modules or related text-messages

INTERVENTIONS:
Behavioral: Personalized feedback — Material includes feedback on alcohol-related consequences with elements from Acceptance Commitment Therapy, Relapse Prevention, Cognitive Behavioral Therapy, and Behavioral Activation. Focus of the intervention is learning about personal environmental cues.
  Other Names: Decisions During Drinking
  Arms: D3 online health information and text-messages

SUMMARY:
Decisions during drinking (D3) is randomized clinical feasibility trial assessing whether health-related materials created for young adults who want to have more positive experiences if they decide to drink alcohol are acceptable and usable. Enrolled participants will be randomized to receive the health-related messages in 5-7 online modules over the 20-30 days or to only receive assessments. Those randomized to receive the intervention will also receive text-messages with health message content during the 20-30 days. After completing the intervention, participants will report on the usability and acceptability of the material, which is the main outcome. For secondary outcomes, participants in both the intervention and control will report on their drinking and drinking-related consequences in the post-intervention questionnaire (or 30 days after initial questionnaire for control participants) and 1 month later.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-24
* At least 1 occurrence of heavy drinking in the past month
* At least 2 alcohol related consequences in the past month
* Live in Washington State
* Agree to be randomized to receive intervention to assessment only control
* Ability to receive SMS text-messages
* Complete Identification verification

Exclusion Criteria:

* Not meeting inclusion criteria
* Not being able to verify identification

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Usability of intervention | From invitation to the first intervention module to end of modules being available 37 days later
  Usability of the intervention is assessed in the intervention group only using a 10-item scale with response options that range from 1 "strongly disagree" to 5 "strongly agree"
Acceptability of the intervention | From invitation to the first intervention module to end of modules being available 37 days later
  Acceptability of the intervention is assessed only in the intervention group using a questionnaire of 11 items each of which is participants will provide as response between 1 "Strongly Disagree" to 7 "Strongly Agree".
Feasibility of intervention | From invitation to the first intervention module to the end of the study 2 months later
  Feasibility will be assessed by the percentage of participants randomized to the intervention that complete the intervention and the 1 month follow-up assessment

SECONDARY OUTCOMES:
Alcohol consumption | From completion of baseline survey to 1 month follow-up approximately 67 days later
  Alcohol consumption will be assessed using the Daily drinking questionnaire, which assesses the number of drinks consumed each day in a typical week in the past month
Alcohol related consequences | From completion of baseline survey to 1 month follow-up approximately 67 days later
  Past month alcohol related consequences will be assessed with 49 questions from several scales including the Rutgers Alcohol Problems Index, Young Adult Alcohol Problems Scale, and the Alcohol-Related Sexual Consequences. All questions except the Alcohol-Related Sexual Consequences are answered on a scale of 0 "Never" to 4 "More than 10 times". Alcohol-Related Sexual Consequences responses are 0 "No" and 1 "Yes" to indicate any occurrence in the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney Hultgren, PhD, Principal Investigator — University of Washington
Locations (1):
- Center for the Study of Health and Risk Behavior, University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to NIAAA data archive (NIAAADA).
Supporting Information: Study Protocol
Time Frame: Data will be uploaded to the NIAAA by October 2025 and be publicly available by September 2028 (two years after the end of data collection).
Access Criteria: To access individual level data researchers need to receive authorization by initiating a Data Access Request (DAR), completing the NDA Data Use Certification (DUC) within the DAR, and satisfying several pre-requisites. DARs will be reviewed by a special committee at NIAAA to ensure that the researcher has provided adequate information for the responsible use of the data per the terms of the DUC. https://nda.nih.gov/niaaa/getting-data-access